CLINICAL TRIAL: NCT05248633
Title: Bortezomib-lenalidomide-dexamethasone Combined With Radiotherapy for Newly Diagnosed Solitary Plasmacytoma
Brief Title: Chemotherapy Combined With Radiotherapy Versus Radiotherapy Alone for Solitary Plasmacytoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SP2022
Record Dates: First submitted 2022-02-18; First posted 2022-02-21 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-06

CONDITIONS: Solitary Plasmacytoma
MeSH Terms: conditions — Neoplasms, Plasma Cell | interventions — Radiotherapy; Bortezomib; Lenalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radiotherapy (Active Comparator)
  Interventions: Radiation: radiotherapy
- Chemotherapy combined with radiotherapy (Experimental)
  Interventions: Radiation: radiotherapy; Drug: Bortezomib Injection; Drug: Lenalidomide; Drug: Dexamethasone

INTERVENTIONS:
Radiation: radiotherapy — radiotherapy with a dose of 40-50 Gy
Drug: Bortezomib Injection — subcutaneous Bortezomib 1.3mg/m2 d1,8,15,22
  Arms: Chemotherapy combined with radiotherapy
Drug: Lenalidomide — Lenalidomide 25mg for 21 days
  Arms: Chemotherapy combined with radiotherapy
Drug: Dexamethasone — Dexamethasone 40mg d1,8,15,22
  Arms: Chemotherapy combined with radiotherapy

SUMMARY:
Solitary plasmacytoma (SP) is characterized by a localized mass of clonal plasma cells with no or minimal bone marrow plasmacytosis. It can present either as EMP or SBP. Radiotherapy is the first-line treatment with high response rate. However, 65-84% SBP patients and 25-35% EMP patients progress at 10 years. We aimed to investigate whether adjuvant bortezomib based chemotherapy with radiotherapy could prolong event-free survival in treatment-naive SP patients compared to that with radiotherapy alone.

ELIGIBILITY:
Inclusion Criteria:

* treatment-naïve SP.

Exclusion Criteria:

* Not appropriate for radiotherapy.
* ECOG > 2.
* Co-morbidity of uncontrolled infection.
* Co-morbidity of other active malignancy.
* Patients in pregnancy or lactation.
* Prior or concurrent pulmonary embolism.
* Patients not able to tolerate thrombosis prophylaxis, bortezomib, lenalidomide or dexamethasone.
* Seropositive for human immunodeficiency virus, seropositive for hepatitis C, or HBV-DNA > 1000 copies/mL.
* Myocardial infarction, NYHA Class III or IV heart failure, uncontrolled angina, severe uncontrolled arrhythmias within 6 months prior to enrollment.
* Grade 2 or higher neuropathy according to National Cancer Institute Common Terminology Criteria for Adverse Events.
* Neutrophil <1×10E9/L，hemoglobin < 8g/dL，or platelet < 75×10E9/L.
* Severely compromised hepatic or renal function: ALT or AST > 3 × ULN, total bilirubin > 1.5 × ULN，or eGFR < 40mL/min.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2022-04-21 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
event-free survival | 2 years
  EFS was calculated from randomization to local progression, local recurrence, distant recurrence, development of smoldering multiple myeloma, multiple myeloma or death.

SECONDARY OUTCOMES:
overall survival | 2 years
  OS was calculated from randomization to death
response rate | 2 years
  assessed according to M protein level, RECIST 1.1 and PET-CT
adverse events | collected until 30 days after treatment completion
  graded according to CTCAE

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, China